CLINICAL TRIAL: NCT05232981
Title: Conservative Management of Placenta Accreta Spectrum With or Without Internal Iliac Ligation: A Randomized Controlled Trial
Brief Title: Conservative Treatment of PAS With or Without IIL
Acronym: PASIIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Assistant professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PASIIL
Record Dates: First submitted 2022-01-28; First posted 2022-02-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Placenta Accreta; Cesarean Hysterectomy; Pelvic Devascularization
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients only will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Conservative management of PAS with Ligation of the bilateral internal iliac arteries
  Interventions: Procedure: Ligation of the bilateral internal iliac arteries
- Control group (Active Comparator): Conservative treatment with Shehata's technique and no internal iliac ligation
  Interventions: Procedure: Shehat's technique

INTERVENTIONS:
Procedure: Ligation of the bilateral internal iliac arteries — opening the posterior peritoneum overlying the bifurcation of the common iliac arteries. Then careful dissection of the internal iliac artery is carried out on each side and the anterior division of the internal iliac artery is ligated 4 cm below the bifurcation of the common iliac on both sides by single ligation procedure using Vicryl 1.0 .
  Re-checking of the femoral pulsation of both sides is performed. Then, the placenta is removed manually in a piecemeal manner, any remaining bleeding points from the placental site are then controlled by hemostatic sutures .
  Arms: Study group
Procedure: Shehat's technique — The three-step technique (Shehata's technique) entailed 3 steps, the first step is double bilateral ligation of uterine arteries before placental separation. Uterine artery ligation is made at 2 levels. First will be done at the isthmus and second will be done 1 cm above the cesarean incision. Regarding timing of ligation , we will apply the uterine artery ligation before placental separation to minimize blood loss at the attempt of placental separation.
  Placenta is separated manually either totally or in piecemeal. If manual separation failed, placenta is removed by scissors.
  Application of quadruple sutures is done at the lower uterine segment to compress and secure the neovascularization in the bed of placenta.
  Insertion of triple way catheter is commenced from inside the uterine incision downwards using long artery forceps or uterine sound and the pulled by the assistant from below. The catheter balloon is inflated by 50 cc saline and left for 48 hours
  Arms: Control group

SUMMARY:
In the current study, the investigators aimed to compare the benefits of internal iliac ligation in placenta accreta spectrum

DETAILED DESCRIPTION:
This randomized control trial will be conducted at Tanta University hospital, Egypt, from 2022 to 2024. Tanta University Hospital is considered the main tertiary hospital at the center of Nile Delta .

Cases, suspected to have PAS, are recruited from the outpatient clinic, and subsequently transferred for ultrasonod gray scale and dopplar for assessment of placental location, invasion and commont on the fetus .

Cases are diagnosed to have PAS by the following criteria Placenta lacunae , Loss of clear zone , Bladder wall interruption, uterovesical hypervascularity and increased vascularity in inferior part of lower uterine segment extending into parametrial region9 will be included in the study. MRI will be done if ultrasonod isn't conclusive , cases with posterior placenta, depth of placental invasion, relationship to posterior bladder wall and presence of parametrial invasion .

All cases will be subjected to the following:

1. A written consent will be obtained from the patients after informing them about the risk of intrapartum and postpartum hemorrhage, the need for blood transfusion, and the possibility of hysterectomy if needed to stop massive blood loss. The consent is approved by the medical ethical committee of Tanta University Hospital.
2. Full history taking with special attention on:

   * Age of the patient .
   * Obstetric History especially number of children and sex .
   * Detailed history of previous deliveries and gynecological procedures.
   * History of any previous surgery.
3. Full general and abdominal examination including weight, height, body mass index (BMI) and blood pressure.
4. Routine lab investigation : CBC, coagulation profile ( PT , PTT , Bleeding time , Clotting time ) , ABO , RH Typing , virology .

Randamisation and Allocation :

Patients will be given aclosed envelope containing either letter C or letter I . The envelope that opened by patient will not change allocation .

The enrolled cases will be allocated into two groups with 1:1 allocation. Group 1 :( Study group ) include cases that will undergo bilateral internal iliac arteries ligation .

Group II :( Control group ) will undergo conservative management by three step technique (Shehata's technique) .

Intervention

Preoperative preparation :

Planned elective CS ≤ 37 wk unless the clinical situations necessitate earlier termination of pregnancy.

A multidisciplinary team including a two senior obstetricians, vascular surgeon , a urologist, an anesthesiologist, and a pediatrician are involved in the operation.

Four units of cross-matched blood are prepared for each patient .Ureteric catheters will be prepared to be used when indicated . Drugs that control bleeding will be preparedsuch as Oxytocin, Carbetocin, Ergometrine, Misoprostol and Tranexamic acid.

All cases undergo general anesthesia by a specialized team. The operation started with Pfannenstiel skin incision and careful dissection of urinary bladder till exposing the uterus.

Uterine incision above placental edge will be done to avoid transplacental incision that triggers heavy bleeding and then extraction of the baby with ecbolic administration, the uterus with the placenta inside will be exteriorized outside the abdomen .Redissecion of U.B will be done if previous dissection at the beginning of the surgery is insuffient.

ELIGIBILITY:
Inclusion Criteria:

1. Age under 35 years old.
2. Prenatally diagnosed placenta accreta .
3. Planned caesarean section ≤ 37 wks .
4. ≤ previous 3 ceserian sections .
5. Placenta accretta spectrum grade 1 , 2 ,3 .
6. Patients who want to preserve their fertility.
7. Patients who refuse hysterectomy .

Exclusion Criteria:

1. Cases with high risk of intraoperative blood loss as hemorrhagic disorders and thrombocytopenia .
2. Cases on anticoagulant therapy.
3. Patients who completed her family.
4. Hemodynamicaly unstable patients.
5. Finally cases who refused to get enrolled in the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | 6 months
  the volume of blood collected in the suction apparatus, excluding the volume of liquor collected, this will be done by meticulous recording of the blood volume in the suction apparatus before opening the uterus and then calculating the exactly added amount of liquor, so that it becomes excluded from the calculation) to the calculated volume of blood obtained from the pre and postoperative difference in weight of the towels and drapes placed beneath the patients, using the following formula: (WET Item Gram Weight - DRY Item Gram Weight¼milliliters of blood within the item) .
Cesarean hysterectomy rate | 6 months
  The success of procedure in prevention of hysterectomy

SECONDARY OUTCOMES:
Operative time | intraoperative
  From skin to skin duration in minutes
Operative and postoperative complications | 6 months
  Any operative organ injury

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Dawood, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
On valuable request
Supporting Information: Study Protocol, SAP
Time Frame: 6 months
Access Criteria: full acess